CLINICAL TRIAL: NCT00479700
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of SAM-531 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAM-531 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3193A1-100
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

INTERVENTIONS:
Drug: SAM-531

SUMMARY:
To assess the safety and tolerability of ascending single oral doses of SAM-531 in healthy subjects.To obtain preliminary pharmacokinetic (PK) and pharmacodynamic (PD) profiles of SAM-531, an investigational drug, in healthy subjects and to evaluate the effect of a high-fat meal on the PK of SAM-531 administered to healthy subjects.

ELIGIBILITY:
Inclusion criteria

1. Men or women of nonchildbearing potential aged 18 to 45 years
2. Elderly men or women aged 65 years and above as of study day 1.
3. Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg. Body weight for elderly subjects must be ≥45 kg.

Exclusion criteria

1. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease
2. Any clinically important deviation from normal limits in physical examination, vital signs, digital 12-lead ECGs, or clinical laboratory test results.
3. Tobacco use or the consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours before study day 1, or grapefruit or grapefruit-containing products 72 hours before study day 1, and until the end of the inpatient confinement period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2006-05; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer